CLINICAL TRIAL: NCT07154342
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of GR1802 Injection in Combination With Background Therapy in Patients With SAR
Brief Title: A Study of IL4Rα Monoclonal Antibody in Patients With Seasonal Allergic Rhinitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-014
Record Dates: First submitted 2025-08-13; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Allergic Rhinitis, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interleukin-4 receptor responder (Experimental)
  Interventions: Biological: GR1802 injection
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GR1802 injection — Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Arms: Interleukin-4 receptor responder
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a non-infectious chronic inflammatory disease of the nasal mucosa mainly mediated by immunoglobulin E after exposure to allergens in atopic individuals. The typical symptoms of AR are paroxysmal sneezing, watery rhinorrhea, itching, and nasal congestion, which may be accompanied by ocular symptoms, including eye itching, tearing, redness, and burning sensation, which are more common in patients with hay fever allergies.

ELIGIBILITY:
Main Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Seasonal allergic rhinitis has been prevalent for at least 2 years.
3. Poor control of seasonal allergic rhinitis with nasal glucocorticoids or other therapeutic agents during the same pollen season in the past.
4. Positive serum-specific IgE test results.
5. Symptom severity scores for the season met the enrollment criteria.

Main Exclusion Criteria:

1. Other nasal comorbidities or co-morbidities/states that may be present at the time of screening that affect efficacy determination.
2. Subjects whose allergen exposures in their home or work environments may be expected to change significantly during the trial period.
3. Subjects with poorly controlled recent asthma conditions.
4. Presence of current or past history of infection of special concern, e.g., active tuberculosis, helminthic infections, severe herpes virus infections, etc.
5. Previous use of anti-interleukin 4 receptor alpha subunit (IL4Rα) monoclonal antibody.
6. Have a serious underlying medical condition that, in the opinion of the investigator, may pose a risk to subject safety by participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in rTNSS( reflective total nasal symptom scores) | up to 2 weeks
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline in rTOSS( reflective total ocular symptom scores) | up to 2、4 weeks
  Scores range from 0 to 9, with higher scores indicating more severe symptoms.
Change from Baseline in rTNSS | up to 4 weeks
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.
Mean change from baseline in iTNSS(instantaneous total nasal symptom scores) | week 2、4
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.
Mean change from baseline in iTOSS(instantaneous total ocular symptom scores) | week 2、4
  Scores range from 0 to 9, with higher scores indicating more severe symptoms.
Change from baseline in RQLQ(Rhinoconjunctivitis Quality of Life Questionnaire) scores | week2、4
  There are 28 questions in 7 fields，Each question is answered on a 7-point scale (0 to 6).
Adverse events (AEs) | up to 12 weeks
Incidence of ADAs | up to 12 weeks
Ctrough | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan university, Wuhan, Hubei, China